CLINICAL TRIAL: NCT06563037
Title: The Effect of Hallux Valgus Angle on Dynamic Knee Movement Pattern
Status: Completed | Type: Observational
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Principal Investigator, Emre Serdar Atalay, Assist. Prof., Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey
Other Study IDs: E-77082166-604.01.02-39435
Record Dates: First submitted 2024-08-11; First posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Hallux Valgus
Keywords: Hallux valgus; Injury; Judo; Knee; Weightlifting
MeSH Terms: conditions — Hallux Valgus; Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Weightlifters and Judo Athletes: At least 3 years of experience in their respective sports. Athletes without acute injuries that could affect performance tests were included.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is an observational study

SUMMARY:
Abstract Background/aim: Little is known about the relationship between hallux valgus and the alignment of proximal joints. Dynamic knee valgus is a movement pattern characterized by excessive knee abduction along with femoral adduction, internal rotation, and relative external tibial rotation. It is more prevalent in females and exacerbates during landing in jumping, predisposing athletes to injuries. The aim of this study is to investigate the effect of hallux valgus deformity on dynamic knee movement pattern and lower extremity injuries in athletes.

Materials and methods: This is a cross-sectional observational study. The study included 92 athletes with at least 3 years of experience in their respective sports.

DETAILED DESCRIPTION:
Athletes without acute injuries that could affect performance tests were included. Demographic data were collected, and the hallux valgus angle was measured using a goniometer. A standard warm-up protocol was then administered. A drop jump test from a 30cm platform was conducted, and images captured during the test were analyzed in 2D using Kistler+Noraxon Measurement Device cameras.

ELIGIBILITY:
Inclusion Criteria:

* At least 3 years of experience in their respective sports.

Exclusion Criteria:

* Athletes with acute injuries

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: At leat 3 years of experienced judo and weightlifters
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2022-06-07 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
Drop Jump Test | 30 minutes
  The drop jump test from a 30cm platform was conducted, and images captured during the test were analyzed in 2D using Kistler+Noraxon Measurement Device cameras. Two cameras were used, one placed in the coronal plane to view the participant from the front, and the other placed in the sagittal plane to view from the left side. Reflective markers were attached to the reference points for measurements

SECONDARY OUTCOMES:
Hallux Valgus Angle Measurement | 10 minutes
  Hallux valgus angle involves measuring the angle between the long axis of the first metatarsal bone and the longitudinal axis of the first phalanx [15]. The normal value ranges from 8˚ to 10˚. However, some authors suggest lateral deviation up to 15˚ may be considered normal

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences Turkey, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hewett TE, Myer GD, Ford KR, Heidt RS Jr, Colosimo AJ, McLean SG, van den Bogert AJ, Paterno MV, Succop P. Biomechanical measures of neuromuscular control and valgus loading of the knee predict anterior cruciate ligament injury risk in female athletes: a prospective study. Am J Sports Med. 2005 Apr;33(4):492-501. doi: 10.1177/0363546504269591. Epub 2005 Feb 8. PMID 15722287